CLINICAL TRIAL: NCT02856282
Title: Drug Utilization Study for Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
Brief Title: Drug Utilization Study for Pirinase Hayfever Relief
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 205708
Record Dates: First submitted 2016-03-24; First posted 2016-08-04 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Nasal Sprays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pirinase Hayfever Relief for Adults 0.05% Nasal Spray: Two sprays into each nostril once a day, preferably in the morning. Once symptoms are under control ,a maintenance dose of one spray may be used accordingly
  Interventions: Drug: Pirinase Hayfever Relief for Adults 0.05% Nasal Spray

INTERVENTIONS:
Drug: Pirinase Hayfever Relief for Adults 0.05% Nasal Spray — Aqueous suspension of 0.05% micronised fluticasone propionate.Each actuation contains 50 micrograms of fluticasone propionate

SUMMARY:
The purpose is to obtain real-world information on how consumers are complying with the product labelling This study will coincide with the launch of Pirinase Hayfever Relief for Adults 0.05% Nasal Spray in the United Kingdom (UK).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be required to review, and electronically sign a Participation Agreement prior to completing the online survey.
* Participants of any age may participate.
* Participants who have purchased and used Pirinase Hayfever Relief for Adults 0.05% Nasal Spray for at least 7 days and are willing to participate in the online survey.
* Participants of either gender may participate

Exclusion Criteria:

* Anyone who is directly involved with medicines such as doctors, nurses, and pharmacists.
* Participants who decline participation in the online survey

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: An all comers population (consumers who opt in at their own discretion) of approximately 1,537 consumers, will be included in this study. Age, gender, and social backgrounds will be allowed to fall out naturally.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Brentford, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in United Kingdom. Participants who purchased product took part in online survey conducted by either of 2 methods: 1- scanned a Quick Response code on product package labelling/link on the product box, 2- via an e-mail invitation (who purchased product at a Boots Pharmacy), that included a link to the survey.
Pre-assignment Details: A total of 72 participants were screened out of whom only 46 answered the survey. Rest 31 were screen failures.
Groups:
- Pirinase Hayfever Relief for Adults 0.05% Nasal Spray: Participants were advised to take Pirinase Hayfever Relief for Adults 0.05 percent (%) Nasal Spray (an aqueous suspension of 0.05% micronised fluticasone propionate), two sprays into each nostril once a day, preferably in the morning for at least 7 days. Participants were invited to complete the online survey if they qualified the screening and were using the product for at least 1 month. Data collection continued through 2 allergy seasons (up to a maximum of 2 years).
Period: Overall Study
Arm/Group | Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
Started | 46
Completed | 45
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included a total of 46 participants who initiated the online survey and no participant was excluded from baseline analysis.
Arm/Group | Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 39
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Used the Test Product at Correct Age (18 Years or Older)
Description: Participants who answered the question, 'What is your age?', were evaluated to provide the data for this outcome measure.
Time Frame: 2 allergy seasons (up to a maximum of 2 years)
Population: Analysis population included all participants who completed the online survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
Number analyzed (Participants) | 45
Participants | 45

2. Primary Outcome: Number of Participants Who Did Not Exceed the Correct Frequency of Use (2 Sprays Per Nostril Per Day)
Description: Participants who answered the question, 'When using Pirinase Hayfever Relief for Adults 0.05% Nasal Spray product, did you use more than 2 sprays in each nostril per day?,' were evaluated to provide the data for this outcome measure.
Time Frame: 2 allergy seasons (up to a maximum of 2 years)
Population: Analysis population included all participants who completed the online survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
Number analyzed (Participants) | 45
Participants | 32

3. Primary Outcome: Number of Participants With Improved Symptoms Who Reduced the Doses to 1 Spray Per Nostril Per Day
Description: Participants who answered the question, 'Did you reduce the dose to 1 dose per nostril after your symptoms improved?', were evaluated to provide the data for this outcome measure.
Time Frame: 2 allergy seasons (up to a maximum of 2 years)
Population: Analysis population included all participants who completed the online survey. Here, number of participants analyzed indicates, participants who answered the question for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
Number analyzed (Participants) | 41
Participants | 30

4. Primary Outcome: Number of Pregnant/ Breastfeeding Participants Who Consulted Physician Before Product Use
Description: Participants who answered the question, 'Did you talk to your doctor before using Pirinase Hayfever Relief for Adults 0.05% Nasal Spray product (if consumer said yes to pregnant or breastfeeding)? ', were evaluated to provide the data for this outcome measure.
Time Frame: 2 allergy seasons (up to a maximum of 2 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
Number analyzed (Participants) | 23
Participants | 0

5. Primary Outcome: Number of Participants Who Consulted Physician if Symptoms Were Not Improved After Using Test Product for 7 Days
Description: Participants who answered the question, 'Did you consult a doctor about your symptoms not improving after using Pirinase Hayfever Relief for Adults 0.05% Nasal Spray product for 7 days? ', were evaluated to provide the data for this outcome measure.
Time Frame: 2 allergy seasons (up to a maximum of 2 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
Number analyzed (Participants) | 4
Participants | 0

6. Secondary Outcome: Number of Participants Who Used the Test Product and Were Not Taking a Medication for Human Immunodeficiency Virus (HIV)
Description: Participants who answered the question, 'Do you take medicine for HIV?', were evaluated to provide the data for this outcome measure.
Time Frame: 2 allergy seasons (up to a maximum of 2 years)
Population: Analysis population included all participants who completed the online survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
Number analyzed (Participants) | 45
Participants | 44

7. Secondary Outcome: Number of Participants Who Consulted Physician When Test Product Was Used for 1 Month or More Continuously
Description: Participants who answered the question, 'Did you consult with a doctor about continuing to use Pirinase Hayfever Relief for Adults 0.05% Nasal Spray product (if consumer answered no to symptoms improving)?', were evaluated to provide the data for this outcome measure.
Time Frame: 2 allergy seasons (up to a maximum of 2 years)
Population: Analysis population included all participants (N=39) who used the test product for atleast 1 month. Here, number of participants analyzed indicates, participants who answered the question for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
Number analyzed (Participants) | 11
Participants | 3

ADVERSE EVENTS:
Time Frame: 2 calendar years from the date of screening
Description: Adverse events were not prompted in this study but a reference to the yellow card scheme for reporting of side effects was included at the end of the survey.
Arm/Group | Pirinase Hayfever Relief for Adults 0.05% Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT02856282/SAP_000.pdf
  • Study Protocol (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT02856282/Prot_001.pdf